CLINICAL TRIAL: NCT00270946
Title: A Pivotal Study to Evaluate the Safety and Efficacy of Cryopreserved Bilayered Cellular Matrix (OrCel) for the Treatment of Venous Ulcers
Brief Title: Evaluation of Bilayered Cellular Matrix (OrCel) for the Treatment of Venous Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ortec International (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100-VLU-01-CLN
Record Dates: First submitted 2005-12-28; First posted 2005-12-29 (Estimated); Last update posted 2005-12-29 (Estimated); Status verified 2005-12

CONDITIONS: Venous Leg Ulcer; Venous Stasis Ulcer
Keywords: Venous leg ulcer; OrCel; Compression therapy
MeSH Terms: conditions — Varicose Ulcer

INTERVENTIONS:
Device: Bilayered Cellular Matrix (OrCel)

SUMMARY:
This study was designed to evaluate the clinical benefits and safety of OrCel in the treatment of venous ulcers. OrCel and standard care were compared to standard care alone. Standard care consisted of currently accepted compression therapy.

Patients were treated for 12 weeks. Patients with healed ulcers were followed for an additional 12 weeks to assess durability of the healed wound.

ELIGIBILITY:
Inclusion Criteria:

* Any race, between 18 and 85 years of age
* Male or female
* Chronic venous insufficiency
* Ulcer size between 2 and 20 sq cm, inclusive
* Ulcer present for at least one month
* ABI >0.7

Exclusion Criteria:

* Decrease in wound size >35% during Screening Phase
* Infection at the ulcer site
* Uncontrolled diabetes mellitus
* Previous treatment with excluded medications

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2002-04; Study Completion 2003-12

PRIMARY OUTCOMES:
Investigator assessment of wound healing

SECONDARY OUTCOMES:
Planimetric assessment of wound healing
Photographic assessment of wound healing

CONTACTS AND LOCATIONS:
Locations (1):
- Terry Treadwell, MD, Montgomery, Alabama, United States